CLINICAL TRIAL: NCT02160106
Title: First-in-Human Dose-Escalation Study of Vactosertib (TEW-7197) Monotherapy in Subjects With Advanced Stage Solid Tumors
Brief Title: First in Human Dose Escalation Study of Vactosertib (TEW-7197) in Subjects With Advanced Stage Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MedPacto, Inc. (Industry)
Collaborators: National OncoVenture (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-001
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2019-05

CONDITIONS: Advanced Stage Solid Tumors
Keywords: Cancer; advanced solid tumors; metastatic; phase I; transforming growth factor beta; TGF-β; first-in-human; TEW-7197; activin receptor-like kinase 5; ALK5; Smad2; Smad3; phospho-Smad; phospho Smad; psmad; serine / threonine kinase inhibitor; pharmacokinetics; MedPacto; National OncoVenture
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Camurati-Engelmann Syndrome; Keratoacanthoma familial | interventions — vactosertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TEW-7197 (Experimental): Dose Escalation of TEW-7197: TEW 7191 tablets will be given once daily (QD) or twice daily (BID) for 5 days followed by 2 days without treatment in 28-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons.
  Interventions: Drug: TEW-7197

INTERVENTIONS:
Drug: TEW-7197 — Single daily doses by oral administration on Days 1, 2, 3, 4, 5, Days 8, 9, 10, 11, 12, Days 15, 16, 17, 18, 19 and Days 22, 23, 24, 25, 26 of each 28 day cycle. Starting dose is 30 mg, with escalation to 60 mg, and subsequent dose escalation using a modified Fibonacci algorithm.
  Other Names: EW-7197; EW7197

SUMMARY:
The phase I dose escalation study will investigate the safety, tolerability, and pharmacokinetics of the TGF-β pathway inhibitor TEW 7197 in subjects with advanced, refractory solid tumors.

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose-escalation, phase I study of TEW-7197 in subjects with advanced solid tumors. The study will investigate the safety, tolerability, and pharmacokinetics of TEW-7197, and will define the maximum tolerated dose (MTD) of TEW-7197 using a 3 + 3 design. An expansion phase at the MTD will identify the recommended phase 2 dose, with an emphasis on subjects with melanoma, breast cancer, hepatocellular carcinoma, and prostate cancer. TEW-7197 is an orally bioavailable small molecule that inhibits protein serine/threonine kinase of activin receptor-like kinase 5 (ALK5) and blocks intracellular signaling of TGF-β by inhibiting the phosphorylation of ALK5 substrates.

ELIGIBILITY:
Inclusion Criteria:

* Advanced stage solid tumors as documented by histological or cytological evidence, with no available approved therapies known to cure metastatic disease or extend survival, and who have received all standard therapy.
* Documented disease progression following prior therapy, as assessed by the Investigator.
* Eastern Cooperative Oncology Group (ECOG) 0 or 1.
* Evaluable or measurable disease as defined by RECIST v1.1 may be enrolled in the dose escalation part; for the dose confirmation part, subjects must have measurable disease by RECIST v1.1 or biomarker for response.
* Males and females ≥ 18 years of age.
* Able to give written informed consent.
* Able to swallow tablets.
* Willing and able to comply with scheduled visits, treatment plans, laboratory tests and procedures.
* Acceptable liver function:

  * Bilirubin ≤ 1.5 times the upper limit of normal (ULN),
  * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the ULN; if liver metastases are present, then ≤ 5 times the ULN is allowed.
* Acceptable renal function:

  *Serum creatinine ≤ 1.5 times the ULN.
* Acceptable hematologic status (without growth factor support or transfusion dependency):

  * Absolute neutrophil count (ANC) ≥ 1,500 cells/μL,
  * Platelet count ≥ 100,000/μL,
  * Hemoglobin ≥ 9.0 g/dL.
* QTc interval calculated according to Fridericia's formula (QTcF = QT/RR0.33; RR = RR interval) of ≤ 450 msec on screening electrocardiogram (ECG).
* Must have a normal ejection fraction (within the reference range of the institution) and no clinically significant valvular dysfunction.
* Must have discontinued cancer treatments, including experimental agents for 28 days or a minimum of 5 half-lives (for any biologics) prior to the start of treatment. Enrollment after exposure levels of a biologic have fallen below an active level as established in the summary basis of approval is acceptable.
* Must have discontinued radiotherapy at least 14 days with resolution of any toxicity to Grade 1 or better prior to the start of treatment.
* A life expectancy of at least 3 months as assessed by the Investigator.
* Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days of the first administration of study drug. For the purpose of this study, female subjects of childbearing potential are defined as all female subjects after puberty unless they are postmenopausal for at least 1 year, or are surgically sterile (hysterectomy or bilateral oophorectomy or tubal ligation).

Exclusion Criteria:

* Elevated Troponin 1 levels at screening or known to have persistently elevated brain natriuretic peptide (BNP).
* Serious pre-existing medical conditions as follows:

  * Myocardial infarction within 6 months prior to screening, or pericardial effusion,
  * History of cardiac or aortic surgery,
  * Serious arrhythmia,
  * Unstable angina pectoris,
  * Congestive heart failure of New York Heart Association class III/IV,
  * Hypertension that is not controlled by standard medication (to 150/90 mmHg or below),
  * Cirrhosis of the liver, Child-Pugh Stage B or C, or history of liver transplant,
  * Severe diabetes that is not currently controlled,
  * Current or history of interstitial pneumonitis,
  * Presence of aneurisms of the ascending aorta or aortic stress.
* Uncontrolled metastatic disease to the brain or central nervous system (CNS).
* Known history of difficulty swallowing, malabsorption or other conditions that may reduce absorption of the product.
* Received prior treatment targeting the signaling pathway of TGF-β.
* Major abnormalities identified by ECG or echocardiogram (ECHO), at the Investigator's discretion.
* Known infection of, or who test positive for, human immunodeficiency virus, hepatitis B virus or hepatitis C virus.
* Active infection requiring systemic antibiotic therapy.
* Known substance abuse or receiving concurrent treatment with non-permitted drugs.
* Female subjects who are breastfeeding, or intend to breastfeed during the duration of the study and for 30 days following the last dose of study drug.
* Known history, or suspected hypersensitivity to any excipients.
* Female subjects must not be pregnant or at risk to become pregnant during the study. Fertile male and female subjects must agree to use an effective barrier method of birth control to avoid pregnancy (for female subjects a double-barrier method of contraception, for male subjects a condom with spermicide) or total abstinence from the time of providing informed consent until 90 days after the last administration of study drug. Use of oral contraceptives is not allowed.
* Any other serious medical condition which in the Investigator's opinion would preclude safe participation in the study.
* Subjects, in the opinion of the Investigator, who are unsuitable to participate in the study.
* Currently using or planning to use:

  * Drugs which are exclusively or primarily eliminated by cytochrome P-450 isozyme 3A4 (CYP)3A4.
  * Drugs which are exclusively or primarily eliminated by UDP glucuronyltransferase 1A1 (UGT)1A1.
  * Drugs which are substrates for the drug transporter multidrug resistance protein 1 (MDR1) have a narrow therapeutic window; or which are strong inhibitors of drug transporter MDR1.
* Any major surgeries within 28 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-07-29 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) based on the number of subjects experiencing at least 1 DLT | 28 days

SECONDARY OUTCOMES:
Dose-dependency of toxicity based on: dose limiting toxicities; frequency, type, grade, and seriousness, and causality of treatment-emergent adverse events, and laboratory assessments. | while undergoing study treatment and up to 30 days after the last dose of TEW-7197

CONTACTS AND LOCATIONS:
Overall Officials: Ilho Ha, PhD, Study Chair — MedPacto, Inc.
Locations (2):
- United States (2):
  - Durham, North Carolina
  - Nashville, Tennessee